CLINICAL TRIAL: NCT04283032
Title: Impact of Magnetic Resonance and Biomarkers for Screening for Prostate Cancer With Different Approaches. Cost-effectiveness Analysis (RMP-BX 2018-01)
Brief Title: Impact of Magnetic Resonance and Biomarkers for Screening for Prostate Cancer. Cost-effectiveness Analysis
Acronym: RMPBX201801
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: InvestigatorUrologyIBSAL (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor-Investigator, InvestigatorUrologyIBSAL, MD, Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León
Organization: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Other Study IDs: PI18/01560
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Establish the Efficacy Between the Four Schemes in Terms of the Aggressiveness of the Tumors According to the Gleason Classification; Establish the Efficacy Between the Four Schemes in Terms of Morbidity Associated With the Technique; Establish the Efficacy Between the Four Schemes in Terms of the Patient's Subjective Perception Regarding Pain and Quality of Life; Establish the Association of the Tumor Biomarker in the Early Detection and Aggressiveness of Tumors; Establish the Possible Interaction Between Biomarkers and Resonance in Different Prostate Biopsy Models to Define Tumor Presence and / or Tumor Aggressiveness; Establish the Possible Relationship Between the Expression Profiles of the microRNAs; Establish if There Are Differences Between Transrectal and Transperineal Prostatic Biopsy Schemes in Both Cases With and Without MRI
Keywords: Prostate Cancer; Biomarkers; PSA; MMPm; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Biomarker [-2] proPSA and PHI, microRNAs: miR-141, miR200C, hasa-miR-200b, miR-187, mir-188-5p, miR196b miR-151-3p, miR375, mir-16, miR25 and lec-7c.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Multiparametric magnetic resonance + transrectal biopsy: The patient underwent a previous multiparametric magnetic resonance (RMmp) and a transrectal biopsy (BPTE)
  Interventions: Procedure: Multiparametric magnetic resonance
- Multiparametric magnetic resonance + transperineal biopsy: The patient underwent a previous multiparametric magnetic resonance (RMmp) and a transperineal biopsy (BPTP)
  Interventions: Procedure: Multiparametric magnetic resonance
- Transrectal biopsy: The patient underwent a transrectal biopsy (BPTE)
- Transperineal biopsy: The patient underwent a transperineal biopsy (BPTP)

INTERVENTIONS:
Procedure: Multiparametric magnetic resonance — MRI uses a powerful magnetic field, pulsed radiofrequency and a computer to create detailed images of organs, soft tissues, bones, and practically the rest of the internal structures of the body. MRI does not use ionizing radiation (X-rays).
  Other Names: Transrectal biopsy; Transperineal biopsy
  Groups: Multiparametric magnetic resonance + transperineal biopsy; Multiparametric magnetic resonance + transrectal biopsy

SUMMARY:
Objectives: To establish if there are differences between an ultrasound-guided transrectal prostate biopsy (BPTE) and a transperineal prostatic biopsy (BPTP) with and without a multiparametric Magnetic Resonance (RMmp) in patients with clinical suspicion of prostate cancer (PC) to first prostatic biopsy in terms of:

1. Rate of detection and diagnosis of prostate cancer.
2. Aggressiveness of the detected tumors.
3. Association of the marker [-2] proPSA and the prostate cancer health index (PHI) and microRNAs for the diagnosis of tumors.
4. Adverse effects of the intervention and subjective perception of the patient: pain and degree of satisfaction, and impairment of quality of life.
5. Cost-effectiveness analysis of the different intervention options.

Study Design: Randomized, single-blind prospective clinical study to compare four schemes: RMmp + BPTE vs. BPTE 12 cylinders vs RMmp + BPTP vs BPTP 12 cylinders.

Study population: Patients with clinical suspicion of prostate cancer with PSA between 3-20 ng / mL and normal or abnormal rectal examination, candidates for a first prostate biopsy.

Research techniques: BPTE standard of 12 cylinders compared to RMmp previous to BPTE vs BPTP of 12 cylinders compared to BPTP with previous RMmp.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent prior to performing any of the specific procedures of the study
* Age between 50 * - 75 years (* 45 years, if family history)
* Patients with clinical suspicion of prostate cancer
* Indication of a first biopsy during the study period.
* Life expectancy greater than 10 years.

Exclusion Criteria:

* Patients previously randomized in the present study.
* Patients submitted prior to a prostate biopsy.
* Patients with a previous diagnosis of prostate cancer and / or previous prostate surgery.
* Patients with a previous episode of acute prostatitis of infectious origin in the 3 months prior to inclusion in the study.
* Patients with an active urinary tract infection and / or any previous pathology of severity in the 3 months prior to inclusion.
* Impossibility of performing transrectal or transperineal biopsy and / or magnetic resonance.
* Patients who have received hormonal treatment prior to androgen blockade in the 6 months prior to inclusion in the study.
* History of other tumors.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected clinical risk of prostate cancer with total PSA values between 3 and 20 ng / mL, free PSA index / total PSA less than 20% and normal or abnormal rectal examination, candidates for a first prostate biopsy
Sampling Method: Probability Sample
Enrollment: 628 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparation between transrectal and transperineal prostatic biopsy with o without Magnetic Resonance | 6 months
  Establish if there are differences between the transrectal and transperineal prostatic biopsy schemes in both cases with and without MRI, in patients with suspected clinical risk of prostate cancer (total PSA between 3 and 20 ng / mL, free PSA index / Total PSA less than 20% and normal or abnormal rectal examination) in terms of efficacy measured by the detection rate and tumor aggressiveness of the tumors detected, complication rates and cost analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Francisco Gómez Veiga, Salamanca, Spain